CLINICAL TRIAL: NCT00978302
Title: A Double Blind, Placebo (Vehicle) and Standard Care Controlled, Randomised, Parallel Group Study to Investigate the Clinical Safety, Toleration, Systemic Pharmacokinetics and Local Pharmacodynamics of Repeated, Escalating Concentrations of Intradermal RN1001 in Healthy Male Subjects.
Brief Title: Safety Study of Repeated, Escalating Doses of Intradermal Avotermin (Juvista)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: John Hutchison, Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RN1001-319-1001
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Cicatrix; Wound Healing
Keywords: Cicatrix; Scar; Wound healing; Avotermin; TGF beta 3; Juvista; RN1001
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human; Ltbp3 protein, zebrafish

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (vehicle) (Placebo Comparator)
  Interventions: Drug: Placebo (vehicle)
- Avotermin (Experimental)
  Interventions: Drug: Avotermin

INTERVENTIONS:
Drug: Avotermin — Intradermal injection, 50ng/100μl/3mm punch biopsy, once at time of biopsy and again 24 h later
  Other Names: RN1001; Juvista; TGFbeta 3
  Arms: Avotermin
Drug: Avotermin — Intradermal injection, 100ng/100μl/3mm punch biopsy, once at time of biopsy and again 24 h later
  Other Names: RN1001; Juvista; TGFbeta 3
  Arms: Avotermin
Drug: Avotermin — Intradermal injection, 500ng/100μl/3mm punch biopsy, once at time of biopsy and again 24 h later
  Other Names: RN1001; Juvista; TGFbeta 3
  Arms: Avotermin
Drug: Avotermin — Intradermal injection, 1000ng/100μl/3mm punch biopsy, once at time of biopsy and again 24 h later
  Other Names: RN1001; Juvista; TGFbeta 3
  Arms: Avotermin
Drug: Avotermin — Intradermal injection, 1μg/100μl/3mm punch biopsy, once at time of biopsy and again 24 h later
  Other Names: RN1001; Juvista; TGFbeta 3
  Arms: Avotermin
Drug: Avotermin — Intradermal injection, 10μg/100μl/3mm punch biopsy, once at time of biopsy and again 24 h later
  Other Names: RN1001; Juvista; TGFbeta 3
  Arms: Avotermin
Drug: Placebo (vehicle) — Intradermal injection at time of biopsy and again 24 h later
  Arms: Placebo (vehicle)

SUMMARY:
The purpose of this study is to determine the safety and local toleration and histological effects of various dose levels of avotermin (Juvista) injected intradermally in healthy male volunteers.

DETAILED DESCRIPTION:
The study was split into two Cohorts: A and B. Volunteers in Cohort A were assigned to one of four dose groups receiving 50, 100, 500 and 1000ng/100μl/3mm punch biopsy. Volunteers were assigned sequentially in order of ascending dose. Within each dose group volunteers were further randomised to subgroup a, b or c. Each subject was set to receive four 3mm punch biopsies, two on each arm, and intradermal injection of avotermin, placebo or nothing (standard care).

On day 0 two 3mm punch biopsies were administered under local anaesthesia to the inner aspect of one arm of each subject following intradermal injection of avotermin, placebo or nothing. The four subjects in subgroup a received avotermin to one punch biopsy and placebo to the other. The four subjects in subgroup b received avotermin to one punch biopsy and standard care only to the other. The one subject in subgroup c was administered with intradermal placebo to one biopsy and standard care only to the other. 24 h later a further application of intradermal avotermin, placebo or nothing was applied.

While arm 1 was used as a study arm, arm 2 was used for safety procedures. Subjects were then randomised to return on Day 3 or 7 for excision of the first two punch biopsies. At the same time two punch biopsies and the same treatment regime was carried out on the second arm. These were dosed again 24 h later and all were excised on Day 10.

After determining safety and toleration of all doses in Cohort A, new subjects were assigned to Cohort B. These were allocated in ascending order to groups that would receive 1, 10, 50 and 100μg/100μl/3mm punch biopsy, following the same procedures that were used for Cohort A. Only after the first three groups reached Day 10 and the safety data was analysed would the final volunteers be recruited to the 100μg group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, caucasian male subjects
* Weight between 60 and 150 kg and a BMI within the permitted range for their height using Quetelet's index (weight (kg)/height (m) squared. The permitted index is between 15-45 kg/m squared
* Subjects who have a previous history of surgery or minor injury and who have not developed any evidence of hypertrophic or keloid scar formation

Exclusion Criteria:

* Subjects with evidence of hypertrophic or keloid scarring
* Subjects with tattoos or previous scars in the biopsy areas
* Subjects with evidence of any past or present clinically significant disease, particularly coagulation disorders, immuno-mediated conditions and skin diseases and allergies such as eczema
* Subjects with a history of clinically significant allergies, especially drug hypersensitivity to lignocaine or allergy to the surgical dressings to be used in this study
* Subjects with any clinically significant abnormality following review of pre-study laboratory data and full physical examination
* Subjects who are taking or have taken any prescribed drug in the three weeks prior to day 0 and in particular topical or systemic steroids, anti-inflammatory and anti-coagulant drugs
* Subjects who drink more than 28 units of alcohol per week
* Subjects who have evidence of drug abuse
* Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B surface antigen.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2001-05; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
To determine the safety and local toleration of various dose levels of avotermin (Juvista) injected intradermally into healthy male volunteers. | Days 0 and 1 and either 3 and 4 or 7 and 8 in addition to Day 10. A single post-trial follow-up was made between days 17-24.

SECONDARY OUTCOMES:
To determine the systemic PK of various dose levels of avotermin (Juvista) injected intradermally. | Days 0 and 1 and either 3 and 4 or 7 and 8, in addition to day 10. A single post-trial follow-up was made between days 17-24.
To determine the histological effects (re-epithelialisation and wound healing) of avotermin (Juvista) injected intradermally. | Days 3, 7 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Davies, Principal Investigator — Renovo
Locations (1):
- Renovo Clinical Trials Unit, Manchester, Manchester, United Kingdom